CLINICAL TRIAL: NCT02318849
Title: Social and Behavioral Interventions to Increase Solid Organ Donation
Brief Title: Online Intervention for ANHPI College Students
Acronym: iDecide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: R39OT26993
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Tissue and Organ Procurement
Keywords: designated organ donor, college students

STUDY DESIGN:
Intervention Model Description: Online educational intervention of choice to be an organ donor was provided to undergraduate students at three universities. The intervention launch at the universities were sequentially initiated, in random order. The design included cross-sectional assessments (unique respondents at each site over time ) as well as longitudinal assessments (same students repeatedly assessed over time).
Who Masked: Participant
Masking Description: Students did not know the schedule for rolling out the intervention by university.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First initiation site (Experimental): University randomized to receive intervention after 1 baseline assessment. Duration of intervention was 3 semesters. This was University of Hawaii at Manoa (UHM).
  Interventions: Behavioral: Web intervention
- Second initiation site (Experimental): University randomized to receive intervention after 3 baseline assessments. Duration of intervention was 2 semesters. This was University of Hawaii at Hilo (UHH).
  Interventions: Behavioral: Web intervention
- Third initiation site (Experimental): University randomized to receive intervention after 5 baseline assessments. Duration of intervention was 2 semesters. This was Hawaii Pacific University (HPU).
  Interventions: Behavioral: Web intervention

INTERVENTIONS:
Behavioral: Web intervention — interactive website using social media and gamification
  Other Names: iDecide Hawaii

SUMMARY:
Taking advantage of college students' frequent use of online technology, including social networking sites (e.g., Instagram a social media site /Facebook a social networking site) and social media sites (e.g., YouTube), the investigators will create an online intervention that leverages this technology to engage and educate Asian, Native Hawaiian, Pacific Islanders (ANHPI)students about a range of topics related to organ donation following death.

DETAILED DESCRIPTION:
Over 56% of the 120,000 critically ill Americans waiting on transplant waiting lists are ethnic minorities. The proportion of ethnic minorities, including Asian, Native Hawaiian, Pacific Islanders (ANHPI), on waiting lists exceeds their representation in the general population. However, few ANHPI adults are designated organ donors (DOD) on their driver's licenses or in a donor registry. ANHPI college students (aged 18-29) also have low DOD rates, particularly Filipinos. Individuals are typically asked about becoming a DOD when renewing a driver's license; but most never think about OD outside of the short-lived Department of Motor Vehicles (DMV) transaction. Knowing someone's status as a DOD on their license can be an influential factor in solidifying a family's feelings about donating a relative's organs after his/her death, if their consent is necessary. Of those who choose DOD status on a license, most will remain one for life. Intervening with drivers before the date of their license renewal can be difficult to arrange; however, opportunities arise when college students turn 21 and want to renew their license in order to remove formatting / colors signifying that the license belongs to an underage minor (< 21 years old).

Taking advantage of college students' frequent use of online technology, including social networking sites (e.g., Instagram a social media site /Facebook a social networking site) and social media sites (e.g., YouTube), the investigators created an online intervention that leveraged this technology to engage and educate ANHPI students about a range of topics related to organ donation (OD). It will also provide culturally sensitive messages tailored to their interest in or wariness of organ donation and reframe students' attitudes about OD and becoming a DOD. Previous internet interventions to encourage college students to become DODs have not included culturally sensitive approaches for ANHPI, who have unique barriers to OD. The cross-sectional design will test the impact of introducing, sequentially, an online intervention tailored to college students at three universities (UH-Manoa, UH-Hilo, and Hawaii Pacific University). The sequence of when the a university received the intervention was randomly determined; thus, the study's design was a cross-sectional design. The goal was to increase DOD rates in college students, particularly ANHPI and encouraging peer discussions/interactions/advocacy about OD.

Effectiveness will be measured by a change over time in the percentage of students who report being a DOD on their license/donor registry (250 students per university measured across 6 time points; thus, the total sample = 4,500). The investigators anticipate a 12% increase in DOD rate in students who are exposed to the intervention. Increases in DOD status will also be tracked via an increase (over normal rates) in the number of new donors aged 18-29 who register as a donor on Hawaii's online donor registry. To make the study website relevant to college students the investigators will include resources useful for assignments in courses (e.g., both in required "general education" courses- including one on "writing skills", and courses on ethics, religion, sociology, and culture/ ethnic studies, etc.) Students and student organizations will participate in contests to win prizes (e.g., for the best 1-minute DOD focused-YouTube video/ Instagram picture, creating a "caption" for a photo on Instagram, and student organizations who compete for group awards). A goal of the intervention will be to reframe OD by engaging altruistic attitudes based on college students' commitment to "green" sustainability efforts (e.g., "go green, recycle yourself"). Innovative culturally sensitive strategies that can engage, educate, and reframe DOD for college students, including those who find it unappealing (i.e., the "ick factor") are clearly needed. The online intervention will saturate online venues (i.e., YouTube, Instagram) visited frequently by college students, and the investigators will use the new concept of "gamification" to turn college students' learning and advocacy ideas surrounding OD/DOD into a game or contest with their peers. This project builds upon Drs. Albright and Feeley's (consultant - Univ. of Buffalo, Dept. of Communications) previous work to encourage adolescents and young adults to become a DOD; thus, the investigators feel well-suited to design, implement, and evaluate the proposed project. The intervention will increase DOD rates in ANHPI students, and thus, increase the number of ethnic minorities who become deceased organ donors now and for years to come.

ELIGIBILITY:
Inclusion Criteria:

* Must be registered undergraduate student at University of Hawaii at Manoa, University of Hawaii at Hilo, or Hawaii Pacific University
* Must be over the age of 18yrs

Exclusion Criteria:

* Not an undergraduate college student at one of the participating university sites

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4827 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Albright, PhD, MPH, Principal Investigator — University of Hawaii
Locations (1):
- Cheryl Albright, PhD, MPH, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross-sectional samples of undergraduate students were recruited for every survey; thus, numbers that completed a baseline or a post-treatment survey differed by site. Surveys prior to the intervention served as baseline data and surveys after initiation served as intervention results. For example, one site (UHM -Manoa) received only one baseline survey; but 6 post-intervention surveys.Thus, it had small baseline sample; but, large post-test sample.
Groups:
- Second Initiation Site: University randomized to receive intervention after 3 baseline assessment. Duration of intervention was 2 semesters. This was University of Hawaii at Hilo (UHH).
- Third Initiation Site: University randomized to receive intervention after 5 baseline assessment. Duration of intervention was 2 semesters. This was Hawaii Pacific University (HPU).
Period: Pre-intervention Cross Sectional Data
Arm/Group | First Initiation Site | Second Initiation Site | Third Initiation Site
Started | 249 (There was 1 pre-intervention (control) assessment in University of Hawaii at Manoa.) | 677 (There were 3 pre-intervention (control) assessments at University of Hawaii at Hilo.) | 1212 (There were 5 pre-intervention (control) assessments at Hawaii Pacific University.)
Completed | 249 | 677 | 1212
Not Completed | 0 | 0 | 0
Period: Post-intervention Cross Sectional Data
Arm/Group | First Initiation Site | Second Initiation Site | Third Initiation Site
Started (These samples are cross-sectional data; thus, the baseline and post-intevention sample sizes are not the same.) | 1234 (There were 6 post-intervention assessments at University of Hawaii at Manoa.) | 735 (There were 4 post-intervention assessments at University of Hawaii at Hilo.) | 720 (There were 4 post-intervention assessments at Hawaii Pacific University.)
Completed | 1234 | 735 | 720
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We collected cross-sectional surveys at all timespoints in this study. When we conducted the first survey at each site we labeled it a "Baseline survey". Recruitment was university-wide for all online surveys. One site(UHM) had only one baseline, while the other two sites had multiple baseline surveys before their intervention started(UHH and HPU). However, demographics are reported for ALL surveys across all time pointt to provide demographics for our total survey samples (see study design)
Groups:
- Total: Total of all reporting groups
Arm/Group | First Initiation Site | Second Initiation Site | Third Initiation Site | Total
Number analyzed (Participants) | 1483 | 1412 | 1932 | 4827
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.78 (0.37) | 22.77 (0.36) | 22.68 (0.27) | 22.43 (0.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1120 | 929 | 1578 | 3627
  Male | 363 | 483 | 354 | 1200
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 161 | 217 | 306 | 684
  Not Hispanic or Latino | 1313 | 1165 | 1597 | 4075
  Unknown or Not Reported | 9 | 30 | 29 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 38 | 70 | 79 | 187
  Asian | 757 | 358 | 671 | 1786
  Native Hawaiian or Other Pacific Islander | 206 | 374 | 199 | 779
  Black or African American | 21 | 25 | 82 | 128
  White | 264 | 388 | 682 | 1334
  More than one race | 169 | 152 | 146 | 467
  Unknown or Not Reported | 28 | 45 | 73 | 146
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1483 | 1412 | 1932 | 4827

OUTCOME MEASURES:

1. Primary Outcome: Donor Status
Description: number of subjects who are designated organ donor on license
Time Frame: 2 years
Population: Undergraduate students who completed surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | First Initiation Site | Second Initiation Site | Third Initiation Site
Number analyzed (Participants) | 1483 | 1412 | 1932
Participants | 748 | 715 | 1030
Statistical Analysis 1: Comparison: First Initiation Site vs Second Initiation Site vs Third Initiation Site; The null hypothesis was that the of number students who report being a donor (or talking to parents about organ donation) both before and after exposure to the intervention would be equivalent. A secondary null hypothesis would be that longer expsosures to the intervention over time would not increase the number who report becoming a donor at the final assessment; Test type: Superiority; p = 0.009, Mixed Models Analysis; The anaylsis was adjusted for student characteristics; Change in percentage = 0.09

2. Primary Outcome: Talk to Peers/Family
Description: number of subjects who report talking to family or peers about choice be organ donor
Time Frame: 2 years
Population: Undergraduate students who completed surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | First Initiation Site | Second Initiation Site | Third Initiation Site
Number analyzed (Participants) | 1483 | 1412 | 1932
Participants | 555 | 563 | 846
Statistical Analysis 1: Comparison: First Initiation Site vs Second Initiation Site vs Third Initiation Site; Test type: Superiority; p > 0.10, Mixed Models Analysis — Calculated; Change in percentage = 0

ADVERSE EVENTS:
Time Frame: up to 18 months for site 1 (UHM) , up to 12 months for sites 2 and 3 (HPU & UHH) (the two time periods represent entire study period for the three sites)
Description: CTCAE
Arm/Group | First Initiation Site | Second Initiation Site | Third Initiation Site
All-Cause Mortality (participants affected / at risk) | 0/1483 | 0/1412 | 0/1932
Serious Adverse Events (participants affected / at risk) | 0/1483 | 0/1412 | 0/1932
Other Adverse Events (participants affected / at risk) | 0/1483 | 0/1412 | 0/1932

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT02318849/Prot_SAP_000.pdf